CLINICAL TRIAL: NCT02393118
Title: Safety and Efficacy of the BrainPort V200 Device in Individuals Blinded by Traumatic Injury
Brief Title: A Study to Evaluate the BrainPort Vision Device in Individuals Blinded by Traumatic Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wicab (Industry)
Collaborators: The Chicago Lighthouse (Other); Lighthouse Guild (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WCB14-492; CDMRP-DM130076 (Other Grant/Funding Number: U.S. Department of Defense)
Record Dates: First submitted 2015-03-02; First posted 2015-03-19 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Blindness
Keywords: Assistive technology; Non-surgical visual prosthetic; sensory substitution; BrainPort; Blindness; Assistive device
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BrainPort V200 Device (Experimental): Single Arm
  Interventions: Device: BrainPort V200 Device

INTERVENTIONS:
Device: BrainPort V200 Device — Training in clinic on use of the device for 2-3 days (10 hours) followed by in-home use for a minimum of 300 minutes per month over 12 months.

SUMMARY:
The BrainPort V200 Device is a wearable, non-surgical, prosthetic device intended for people who are profoundly blind. The BrainPort V200 translates images captured by a digital camera into electro-tactile stimulation presented on the user's tongue to perceive shape, size, location, and motion of objects within the environment. The purpose of this study is to evaluate the safety and functional performance of the BrainPort V200 device in individuals who have been medically documented as blind, light perception or worse, due to a traumatic injury (cortical or ocular).

ELIGIBILITY:
Inclusion Criteria:

1. A minimum age of 18 years at enrollment.
2. A documented vision diagnosis of light perception or worse bilaterally.
3. Blinded by traumatic injury (i.e., ocular or cortical trauma).
4. Minimum post 12 months diagnosis of blindness.
5. Previous completion of conventional rehabilitation such as orientation and mobility training with a cane or guide dog.
6. Ability to read (or have read to them) and understand study documents and procedures.
7. Ability to provide valid feedback regarding use of the BrainPort device.
8. Access to an accessible computer and internet connection.
9. Willing and able to complete all questionnaires, telephone conferences, device training, and study procedures required by the protocol, after completing an orientation period with the device.
10. Ability to operate a tablet computer.

Exclusion Criteria:

1. Current oral health problems determined by the participant's medical history and an examination of the oral cavity performed by study personnel.
2. History of injury to the tongue resulting in impaired sensation of use of the tongue.
3. Visible open lesions, cold sores, abrasions, blisters, or rash on the tongue, numbness or lack of feeling of the tongue.
4. Piercings on the tongue.
5. Recent or planned oral surgery and/or dental work in the past three months (does not include routine dental health exams/cleanings).
6. Known neuropathies of the tongue or tactile system.
7. History of seizures or epilepsy.
8. If female, pregnant or breast feeding by self-report. Women of child bearing potential must agree to use appropriate birth control to prevent pregnancy for the duration of the study.
9. People with implanted medical devices (i.e., pacemaker, deep brain stimulator, cochlear implant).
10. Any hearing impairments which prevents hearing the device announcements.
11. Any cognitive disabilities (such as Alzheimer's disease), as determined by medical history and/or the Telephone Inventory Cognitive Screening (TICS).
12. Participation in any other clinical trial or research while my confound results in either study.
13. Known allergy to nickel, gold, or any component of stainless steel.
14. Any medical condition that would interfere with performance on the assessments.
15. The Site Principal Investigator does not deem the candidate to be suitable for the study for other reasons not listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of electrical stimulation on the tongue (to demonstrate no occurrence of a clinically significant device-related adverse event) | 12 months
  The primary safety objective is to demonstrate no occurrence of a clinically significant device-related adverse event.
To assess the efficacy of the BrainPort device as measured by an object recognition task (to demonstrate at least 35% of subjects achieve a success rate in object recognition exceeding that expected by chance alone) | 12 months
  The primary efficacy objective is to demonstrate that at least 35% of subjects achieve a success rate in object recognition exceeding that expected by chance alone.

OTHER OUTCOMES:
Text identification task | 12 months
  Words or sequence of numbers will be presented on flashcards and a mobile tablet, subjects will be asked to verbally identify which word or number is presented.
Navigation task | 12 months
  Subjects will be required to identify key characteristics of a room, such as the number of windows and doorways and complete navigation tasks such as following a line, avoiding obstacles, and walking through a doorway without touching any walls.
Change in the effect of assistive technology on perceived quality of life after using the device for one year as measured by the Psychosocial Impact of Assistive Devices Scale (PIADS). | Baseline, 12 months after device training.
Change in self-efficacy after using the device for one year as measured by the General Self-Efficacy Scale (GSES) | Basline, 12 months after device training.
Change in perceived general pain after using the device for one year as measured by the Universal Pain Assessment Tool | Baseline,12 months after device training
Change in satisfaction of the device after using the device for one year, as measured by the Device Satisfaction Survey | One month after start of home use, 12 months after device training
Optional focus group to assess year long experience with the device. | 12 months after device training

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Grant, M.S., Principal Investigator — Wicab, Inc.
Locations (3):
- United States (3):
  - The Chicago Lighthouse for People Who Are Blind or Visually Impaired, Chicago, Illinois
  - Lighthouse Guild, New York, New York
  - Wicab, Inc., Middleton, Wisconsin

REFERENCES:
- [Derived] Grant P, Maeng M, Arango T, Hogle R, Szlyk J, Seiple W. Performance of Real-world Functional Tasks Using an Updated Oral Electronic Vision Device in Persons Blinded by Trauma. Optom Vis Sci. 2018 Sep;95(9):766-773. doi: 10.1097/OPX.0000000000001273. PMID 30169354